CLINICAL TRIAL: NCT01631032
Title: Phase 3 Study of Qi-tonifying Chinese Herbal Products for Treatment of Allergic Rhinitis
Brief Title: Effect of Qi-tonifying Chinese Herbal Products for Treatment of Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Committee on Chinese Medicine and Pharmacy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMRPD1B0081
Record Dates: First submitted 2012-06-17; First posted 2012-06-28 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Chinese herbal products; Qi deficiency
MeSH Terms: conditions — Rhinitis, Allergic | interventions — bu-zhong-yi-qi-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): control group receive placebo capsule with same look, smell and flavor compared with experiment group. The scheme for medication is 3 times a day, 3gm each time, total 9gm per day.
- Chinese herbal products (CHP) (Experimental): CHP group receive Qi-tonifying Chinese herbal products capsule, 3 times a day, 3gm each time, total 9gm per day
  Interventions: Drug: Qi-tonifying Chinese herbal products

INTERVENTIONS:
Drug: Qi-tonifying Chinese herbal products — Chinese herbal products in capsule, 3 times a day, 3gm (6PC of 500mg capsule) each time, total 9gm per day
  Other Names: Bu Zhong Yi Qi Tang; Hochu-ekki-to
  Arms: Chinese herbal products (CHP)

SUMMARY:
Allergic rhinitis is a common but complicated immunologic disorder disease and multiple western medicine has been used for symptom control. Chinese herbal medicine, one of the most commonly used complementary and alternative medicine in Taiwan, has also be used for allergic rhinitis control. This study is designed to explore the efficacy and possible underlying immune-modulation effect of the BZYQT, which is one of the most famous Chinese herbal medicine used for allergic rhinitis in daily practice.

DETAILED DESCRIPTION:
Allergic rhinitis is the type I hypersensitivity reaction of nasal mucosa to environmental allergen. It is characterized by one or more symptoms including sneezing, itching , rhinorrhea and nasal congestion. The prevalence of allergic rhinitis in Taiwan is approximately 20%-30% and increases annually. However, symptom relapse still bothered the majority of patients though there were certain advances in western medicine. In addition, side effects of western medicine, such as lethargy, mouth dryness after taking anti-histamine and immunosuppression after using steroid are also concerned by patient.

Traditional Chinese medicine has been used widely in Taiwan for several disease, especially allergic diseases, such as allergic rhinitis. Among all Chinese herbal products, qi-tonifying regimen play a central role for allergic diseases control. Bu-zhong-yi-qi-tang (BZYQT), one of the famous qi-tonifying herbal products, has been proved to have immuno-modulation effect in previous studies. However, proof of clinical investigation of therapeutic efficacy and cellular level response are still lacking.

In this study, a double-blinded, randomized, placebo control design is applied and total 120 intermittent allergic rhinitis patients will be enrolled in our study. All subjects will be divided into BZYQT and placebo control groups, each group will have 60 subjects. Subjects of BZYQT group will receive capsule of BZYQT, 3gm tid, 9gm a day, while control group will receive similar placebo capsule with same scheme. Total 2 month treatment course will be done. Clinical evaluation, including symptom severity, quality of life and chronic fatigue degree will be done once per month and one month after completed treatment. Additionally, various parameters for immunologic response will be checked before and after the treatment, including the total IgE amount, the ratio of CD4/CD8 of T lymphocytes, the profile of cytokine such as IL-4,IL-5,IL-8,IL-10,IL-13, IFN-γ as well as PGE2, LTC4, sICAM-1 , the mRNA expression of COX2 and neutrophil phagocytosis. Dendritic cell function, presumably the most important immune-response inducer, will also be checked through test for IL-10 and IL-12.

Results will be analyzed statistically including gender analysis. We hope that therapeutic efficacy and possible cellular mechanism of immune-modulation will be elucidated after completing this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more following symptoms: nose itching, sneezing, rhinorrhea with clear nasal discharge, stuffy nose.
* exacerbation times less than 4 days a week or consecutive episodes less than four weeks
* Mite allergy confirmed by Childhood Allergy Panel (CAP)

Exclusion Criteria:

* Use of steroid, antihistamine, Montelukast or other immuno-modulation drugs or duration of drug discontinuation less than one month
* Active infection, including sinusitis
* Vasomotor rhinitis
* Unable to swallow capsule or history of poor medication compliance
* Major organ dysfunction with relevant impaired physical performance status

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in symptom severity at 3 months | Assessment of symptom severity on starting day (day 0), once a month during treatment course (day 30 and day 60), and 1 month after completed treatment (day 90)
  Okuda scoring system for allergic rhinitis severity, Short-form 36 (SF-36) for life quality, visual analogue scale for fatigue severity

SECONDARY OUTCOMES:
Change from Baseline in immunologic biomarkers at 3 months | Laboratory examination on starting day (day 0), once a month during treatment course (day 30 and day 60)
  immunologic biomarker assessment includes: CD4/CD8 count and ratio, relative cytokines of T Cell, activator mediator of PMNs and phargocytosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sien-hung Yang, Ph.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Yang SH, Hong CY, Yu CL. Decreased serum IgE level, decreased IFN-gamma and IL-5 but increased IL-10 production, and suppressed cyclooxygenase 2 mRNA expression in patients with perennial allergic rhinitis after treatment with a new mixed formula of Chinese herbs. Int Immunopharmacol. 2001 Jun;1(6):1173-82. doi: 10.1016/s1567-5769(01)00051-0. PMID 11407311
- [Background] Yang SH, Hong CY, Yu CL. The stimulatory effects of nasal discharge from patients with perennial allergic rhinitis on normal human neutrophils are normalized after treatment with a new mixed formula of Chinese herbs. Int Immunopharmacol. 2002 Nov;2(12):1627-39. doi: 10.1016/s1567-5769(02)00133-9. PMID 12469937
- [Background] Yang SH, Yu CL. Antiinflammatory effects of Bu-zhong-yi-qi-tang in patients with perennial allergic rhinitis. J Ethnopharmacol. 2008 Jan 4;115(1):104-9. doi: 10.1016/j.jep.2007.09.011. Epub 2007 Sep 19. PMID 17980528
- [Background] Yang SH, Yu CL, Chen YL, Chiao SL, Chen ML. Traditional Chinese medicine, Xin-yi-san, reduces nasal symptoms of patients with perennial allergic rhinitis by its diverse immunomodulatory effects. Int Immunopharmacol. 2010 Aug;10(8):951-8. doi: 10.1016/j.intimp.2010.05.008. Epub 2010 May 28. PMID 20546945
- [Background] Fokkens WJ. Antigen-presenting cells in nasal allergy. Allergy. 1999 Nov;54(11):1130-41. doi: 10.1034/j.1398-9995.1999.00104.x. No abstract available. PMID 10604548